CLINICAL TRIAL: NCT03207334
Title: A Phase II, Open-Label Clinical Efficacy Study Defining Genomic Signatures That Correlate With Midostaurin Response in Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: iCare4: Genomic Signatures With Midostaurin in Acute Myeloid Leukemia (UF-HEM-004)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: University of Florida (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-HEM-004; CPKC412AUS61T (Other Grant/Funding Number: Novartis Pharmaceuticals Corporation); IRB201701934 (Other: Univeristy of Florida)
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; genomic signatures; midostaurin; relapsed; refractory; PKC412
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — midostaurin; Cytarabine

STUDY DESIGN:
Intervention Model Description: All patients will receive midostaurin and cytarabine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Midostaurin and Cytarabine (Experimental): Treatment will consist of 3 phases: induction (a 28-42 day cycle), followed by consolidation (up to 4 cycles). Each cycle in the consolidation phase will last 28 days. Subjects will proceed from one phase to the next if they have achieved or maintained a complete remission or complete remission with incomplete blood count recovery by International Working Group 2003 response criteria. Patients may receive a allogeneic hematopoietic stem cell transplant between the end of the induction phase.
  Interventions: Drug: Midostaurin; Drug: Cytarabine

INTERVENTIONS:
Drug: Midostaurin — Induction Phase: 50 mg orally twice daily beginning on day 7 and ending 48 hours prior to beginning the consolidation phase
  Consolidation Phase: 50 mg orally twice daily beginning on Day 6 and ending 48 hours prior to either the start of the next cycle or beginning conditioning therapy for allogenic stem cell transplant.
  Other Names: PKC412; Rydapt
Drug: Cytarabine — Induction Phase: 3 g/m2 (patients 18-65 years old) or 1 g/m2 (patients > 65 years old or those with co-morbidities precluding a higher dose) by vein over 3 hours every 12 hours on Days 1-6.
  Consolidation Phase: 3 g/m2 (patients 18-65 years old) or 1 g/m2 (patients > 65 years old or those with co-morbidities precluding a higher dose) by vein over 3 hours every 12 hours on Days 1, 3, and 5 of each cycle.
  Other Names: Depocyt

SUMMARY:
This is an open label, single arm study of midostaurin in patients with relapsed or refractory AML.

DETAILED DESCRIPTION:
Clinical trials have shown that the multi-kinase inhibitor midostaurin improves survival in patients with AML. The main objective of this study is to investigate its effect (in conjunction with cytarabine) on progression free survival, as well as overall survival and morphologic response rate in patients with relapsed or refractory AML. This study will also attempt to identify specific populations of patients with relapsed or refractory AML who best respond to treatment with midostaurin to enhance treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject prior to registration on the study and the ability for the subject to adhere to the study visit schedule and all the study-related procedures.
* A diagnosis of relapsed or refractory AML. For the purpose of this study, refractory AML is defined as failure to achieve CR after one cycle of induction chemotherapy and relapsed AML is defined as any evidence of disease recurrence after achieving CR of any duration.
* Both males and females ≥ eighteen years of age
* Karnofsky Performance Status of ≥ 70% or Eastern Cooperative Oncology Group (ECOG) performance status < 2 (unless poor performance status is related to the disease).
* Adequate organ function defined as:
* AST and ALT < 2.5 times the upper limit of normal (ULN),
* Serum bilirubin < 2.5 x ULN, and
* Serum creatinine < 1.5 mg/dL or creatinine clearance > 50 mL/min.
* Laboratory values can be outside of this range if secondary to AML disease.
* An ejection fraction of > 45% confirmed by echocardiogram.
* Life expectancy of greater than one month.
* Subjects who previously received midostaurin are allowed if the last dose of midostaurin was given ≥ six months prior to disease relapse.
* Females who are non-pregnant and non-nursing.
* Females of reproductive age and males must agree to avoid getting pregnant or to father a child while on therapy and for five months after the last dose of chemotherapy.
* Women of child-bearing potential (WOCBP) must either agree to continued abstinence from heterosexual intercourse or begin one of the following acceptable methods of birth control: IUD, tubal ligation, or partner must use a latex condom during any sexual contact, even if the partner has undergone a successful vasectomy. Hormonal contraception is an inadequate method of birth control.
* Males must use a latex condom during any sexual contact with WOCBP, even if they have undergone a successful vasectomy (while on therapy and for five months after the last dose of chemotherapy)

Exclusion Criteria:

* Age ≥ of seventy-six years.
* Subjects with the inability to swallow oral medications.
* Clinical evidence of active CNS leukemia.
* A medical history of receiving an allogeneic hematopoietic stem cell transplantation (HSCT).
* Subjects must not have any uncontrolled or intercurrent illness including, but not limited to,
* ongoing or active infection,
* symptomatic congestive heart failure,
* unstable angina pectoris,
* cardiac arrhythmia,
* myocardial infarction within three months,
* poorly controlled hypertension,
* uncontrolled diabetes, or psychiatric illness/social situation that would limit compliance with protocol requirements.
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least five months after the last dose of chemotherapy.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PKC412.
* Previous therapy with midostaurin within six months prior to relapse.
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects demonstrating an inability to comply with the study and/or follow-up procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Up to 6 months
  Compare the progression free survival of patients receiving midostaurin and cytarabine to that historically achieved in patients receiving cytarabine alone

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by National Cancer Institute (NCI) Common Terminology for Adverse Events(CTCAE) v4.0 | Up to 2.5 years
  Assess the incidence and severity of toxicities of midostaurin and cytarabine using CTCAE v4.0
Overall survival | Up to 3.5 years
  Compare the overall survival of patients receiving midostaurin and cytarabine to that historically achieved in patients receiving cytarabine alone
Morphologic response rate | Up to 6 months
  Compare the morphologic response rate (using International Working Group 2003 criteria) of patients receiving midostaurin and cytarabine to that historically achieved in patients receiving cytarabine alone

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Norkin, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No